CLINICAL TRIAL: NCT01728649
Title: Phase 2 Study of Mild Hypothermia in Combination With Acute Cerebral Vascular Reperfusion in the Setting of Acute Ischemic Stroke
Brief Title: Reperfusion With Cooling in Cerebral Acute Ischemia II
Acronym: ReCCLAIM II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to be funded
Sponsor: WellStar Health System (Other)
Responsible Party: Principal Investigator, Dr. Christopher Horn, Assistant Professor of Neurology and Neurosurgery, WellStar Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSNC 02
Record Dates: First submitted 2012-09-05; First posted 2012-11-20 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Ischemic Stroke; Hypothermia
Keywords: Acute Ischemic Stroke; Mild Hypothermia; Stroke; Hypothermia
MeSH Terms: conditions — Ischemic Stroke; Hypothermia; Stroke | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normothermia (No Intervention): As part of standard of care, an interventional reperfusion procedure will be performed on all subjects using current FDA approved devices. After which patient will be started on normothermia attempting to keep core body temp between 38 and 36.5 degrees centigrade. Patients will also undergo blood draws for biomarkers before reperfusion is achieved the immediately, 6 hours then 24 hours after reperfusion.
- Mild Hypothermia (Experimental): As part of standard of care, an interventional reperfusion procedure will be performed on all subjects using current FDA cleared device. Patient will also have a Quattro catheter placed in the femoral vein and temperature brought to 33 degrees centigrade as quickly as possible. They will stay in mild hypothermia for 12 hours and then be rewarmed very slowly. Patients will also undergo blood draws for biomarkers before reperfusion is achieved the immediately, 6 hours then 24 hours after reperfusion.
  Interventions: Other: Mild Hypothermia

INTERVENTIONS:
Other: Mild Hypothermia — Hypothermia will be achieved using the Zoll Thermoguard XP technology with the Quattro catheter. This catheter has a 9.3 Fr diameter and is 4 3cm long. It will be placed in the patients femoral vein via Seldinger technique, before reperfusion is achieved. Hypothermia will be initiated prior to reperfusion. Once temperature has reached 33.5 degrees centigrade the patient will remain at that temperature for 12 hours after which the patient will undergo active gradual rewarming at 0.2 degrees centigrade per hour.
  Other Names: Hypothermia; Therapeutic Hypothermia
  Arms: Mild Hypothermia

SUMMARY:
The purpose of this study is to determine whether reducing a patients body temperature (mild hypothermia of 33 degrees Centigrade) will significantly reduce the risk of brain injury (notably reperfusion injury and hemorrhagic conversion) in patients that have suffered a significant interruption of blood flow to an area of brain (occlusion of large proximal cerebral artery) and have undergone successful removal of that interruption (revascularization).This will be achieved by comparing patients that have undergone hypothermia to those that have not.

DETAILED DESCRIPTION:
This study is designed to examine the safety and proof of concept of therapeutic hypothermia prior to conventional revascularization in subjects experiencing acute ischemic stroke by comparing the results to subjects who remain at normal body temperature (normothermic) and proceed directly to reperfusion via conventional reperfusion intervention. The investigational plan also examines the following outcomes in 85 subjects randomized to either hypothermia or normothermia:

* Regulation of biomarkers indicative of ischemia-reperfusion injury
* Changes in blood brain injury using the Hyperintense Acute Reperfusion Marker (HARM) protocol MRI as a surrogate imaging biomarker
* Incidence of hemorrhagic conversion post reperfusion
* Neurologic function at 90 days post acute ischemic stroke. The results of this study will be used to power a definitive phase III clinical trial evaluating the combination of hypothermia and revascularization versus reperfusion alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any ethnicity and age >/=18 but </= 85 years;
* Symptom onset </=8 hours;
* Symptoms consistent with an ischemic stroke with a large vessel occlusion (Middle Cerebral Artery (MCA), Internal Carotid Artery (ICA) terminus) as determined by vascular imaging, CT or MRI;
* Alberta Stroke Program Early CT Score (ASPECTS) of 5-10 on non-contrast CT of the brain;
* Ability to undergo endovascular reperfusion therapy;
* No contraindications to general anesthesia or allergies to any components associated with the anticipated diagnostic or treatment procedures that cannot be treated;
* A pre-treatment modified Rankin Scale (mRS) of 0 or 1;
* Arterial puncture performed under 8 hours from symptom onset or last seen normal
* Baseline MRI or CT scan shows no hemorrhage;
* National Institutes of Health Stroke Scale (NIHSS) 14-29;
* Subject has either 1) failed iv tissue plasminogen activator (tPA) therapy or 2) contradicted for iv tPA therapy;
* Subject is capable of complying with study procedures and agrees to complete all required study procedures, study visits and associated activities.
* Subject must be able to understand and give written informed consent.

Exclusion Criteria:

* Females of childbearing potential who are pregnant or not using adequate contraception;
* Bleeding diathesis with a platelet count < 50,000 or International Normalized Ratio (INR) >1.5 or any active or recent (within 10 to 30 days) hemorrhage;
* History of genetically confirmed hypercoagulable syndrome;
* Any condition that excludes MRI imaging;
* History of dementia, currently on Aricept or Namenda, or other Alzheimer's like symptoms;
* End stage renal disease on hemodialysis;
* History of cardiac arrest;
* Presence of an inferior vena cava (IVC) filter;
* Contrast dye allergy with history of anaphylaxis, known serious sensitivity to contrast agents or any condition in which angiography is contraindicated;
* Known allergy to meperidine or buspar;
* Sustained hypertension (systolic blood pressure (SBP) > 185 or diastolic blood pressure (DBP) > 110 refractory to treatment);
* Baseline CT/MRI of head showing evidence of mass effect with mid-line shift, hemorrhage, intracranial tumor, arterial vasculitis or dissection, or bilateral stroke;
* Presence of any other serious comorbidity that would be likely to impact life expectancy to less than 6 months or limit subject cooperation or study compliance;
* Concurrent participation in an investigational clinical study that has not completed the follow-up period or planned participation in another study within the next 3 months;
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete, good quality data or the completion of the research study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 90 days
  Evaluation and determination of the following complications pneumonias, central line infections, intra-cerebral hemorrhages, systemic hemorrhages, transient cerebral ischemia, and new strokes.

SECONDARY OUTCOMES:
Hyperintense Acute Reperfusion Marker (HARM) | 48+/- 24 hours
  HARM is a MRI sequence looking at gadolinium enhancement on FLAIR MRI imaging.
Hemorrhagic Conversion | 48hrs
  Acute bleeding into the area of the original stroke based on CT or MRI of the head.
National Institutes of Health Stroke Scale (NIHSS) | 90 days
  NIHSS is a scale from 1-42 to evaluate stroke severity
Modified Rankin Scale (mRS) | 90 days
  mRS is a straightforward evaluation of the functional limitations from stroke
Biomarkers | Before therapy then immediately after, 8hrs, and 24hrs after reperfusion
  These biomarkers are indicative of ischemia-reperfusion injury

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Horn, MD, Principal Investigator — Emory University; Rishi Gupta, MD, Study Director — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States